CLINICAL TRIAL: NCT00022633
Title: Protocol for Assessment of Gemcitabine and Paclitaxel for Metastatic Urothelial Cancer in Patients Aged 70 Years or Older (and in a Cohort of Patients Younger Than 60 Years)
Brief Title: S0028, Gemcitabine and Paclitaxel in Treating Patients With Advanced or Recurrent Cancer of the Urinary Tract
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Permanently Closed Due to Poor Accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068837; S0028 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: recurrent bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; squamous cell carcinoma of the bladder; adenocarcinoma of the bladder; recurrent urethral cancer; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine, paclitaxel (Experimental)
  Interventions: Drug: gemcitabine hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: paclitaxel
  Other Names: Taxol

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine and paclitaxel in treating patients who have advanced or recurrent cancer of the urinary tract.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of enrolling patients aged 70 years and older with advanced or recurrent urothelial cancer to a structured phase II study.
* Determine the anticancer efficacy of gemcitabine and paclitaxel, in terms of objective response rate and 2-year survival, in these elderly patients.
* Assess the toxicity and tolerability of this regimen in these elderly patients.
* Determine the feasibility of using standardized self-report measures of comorbidity, depression, and functional status in these patients.
* Determine the pharmacokinetics of this regimen in these elderly patients and validate this data against similar parameters in patients aged under 60 years.

OUTLINE: This is a multicenter study. Patients are stratified according to age (70 and over vs under 60).

Patients receive paclitaxel IV over 3 hours on day 1 and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 80 patients (60 age 70 and over and 20 under age 60) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed urothelial cancer

  * Transitional cell carcinoma, adenocarcinoma, or squamous carcinoma (bladder, renal pelvis, ureter, or urethra)
* Previously untreated metastatic or locoregionally advanced (i.e., bulky pelvic nodes) disease OR
* Locally recurrent carcinoma after radiotherapy or cystectomy and no longer eligible for further radiotherapy or surgery
* Measurable disease

PATIENT CHARACTERISTICS:

Age:

* 70 and over OR
* Under 60

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* Aspartate aminotransferase (SGOT) or alanine aminotransferase (SGPT) no greater than 2 times ULN

Renal:

* Creatinine no greater than ULN

Other:

* HIV negative
* No other concurrent life-threatening medical disorder that would preclude study participation
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior adjuvant chemotherapy is allowed provided administered more than 10 years ago
* No prior gemcitabine, taxanes, or platinum-based adjuvant chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 28 days since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics
* At least 28 days since prior surgery and recovered

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2001-07; Primary Completion 2008-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Raghavan, MD, PhD, FRACP, FACP, Study Chair — The Cleveland Clinic
Locations (92):
- United States (92):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Clinic of Dr. Judy L. Schmidt, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - AnMed Health Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The purpose of the subset of patients who aged 60 years or younger was to serve as a younger reference group for the pharmacokinetic parameter estimation. Therefore, this younger cohort is not included in analyses of adverse event, efficacy, and feasibility assessment of patient-reported outcome measures.
Groups:
- Paclitaxel + Gemcitabine (Elderly Cohort: Age >= 70); Paclitaxel + Gemcitabine (Younger Cohort: Age < 60): Patients received 1000 mg /m^2 of gemcitabine on Day 1 and 8 and 175 mg/m^2 of paclitaxel on Day 1 intravenously every 21 days for 6 cycles ( 1 cycle = 21 days)
Period: Overall Study
Arm/Group | Paclitaxel + Gemcitabine (Elderly Cohort: Age >= 70) | Paclitaxel + Gemcitabine (Younger Cohort: Age < 60)
Started | 55 | 10
Eligible | 51 | 10
Completed | 23 | 5
Not Completed | 32 | 5
Not completed — Adverse Event | 11 | 1
Not completed — Refusal unrelated to adverse event | 1 | 0
Not completed — Progression/relapse | 9 | 2
Not completed — Death | 4 | 0
Not completed — Other - not protocol specified | 3 | 2
Not completed — Ineligible | 4 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients who started treatment were included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel + Gemcitabine (Elderly Cohort: Age >= 70) | Paclitaxel + Gemcitabine (Younger Cohort: Age < 60) | Total
Number analyzed (Participants) | 51 | 10 | 61
Age, Continuous [Median (Full Range); unit: years] | 76.1 [70.1 to 85.2] | 53.8 [31.2 to 59.7] | 74.6 [31.2 to 85.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 18
  Male | 37 | 6 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 47 | 9 | 56
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 1 | 5
  White | 46 | 7 | 53
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Overall Confirmed Response Rate in the Patients Age 70 and Older (Complete and Partial Response)
Description: Complete response (CR) is defined as complete disappearance of all measurable and non-measurable disease. No new lesions. No disease related symptoms. Partial response (PR) applies only to patients with least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions.
Time Frame: every week for the first 4 weeks and then every 3 weeks for up to 19 weeks
Population: Eligible patients aged 70 years and older who had received any treatment were included in the analysis. Patients aged 60 years or younger who served as a younger reference group for the pharmacokinetic study were excluded from analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel + Gemcitabine (Elderly Cohort: Age >= 70)
Number analyzed (Participants) | 51
percentage of participants | 22 [11 to 35]

2. Secondary Outcome: Progression-free Survival in Patients Aged 70 Years and Older
Description: Measured form date of registration to date of first observation of progression disease, death due to any cause, symptomatic deterioration, or early discontinuation of treatment.
Time Frame: 0-5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Gemcitabine (Elderly Cohort: Age >= 70)
Number analyzed (Participants) | 51
months | 6 [4 to 7]

3. Secondary Outcome: Overall Survival (OS) in Patients Aged 70 Years and Older
Description: Measured from date of registration to date of death due to any cause.
Time Frame: 0-5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Gemcitabine (Elderly Cohort: Age >= 70)
Number analyzed (Participants) | 51
months | 11 [8 to 13]

4. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 2.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Patients were assessed for adverse events weekly after protocol treatment for cycle 1 (1 cycle = 21 days) and then weekly for the first 2 weeks of protocol treatment for cycle 2-6 and after completion of protocol treatment.
Population: Eligible patients aged 70 years and older who had received any treatment were included in the adverse event summaries. Any CTCAE 2.0 event of Grade 3, Grade 4, or Grade 5 which deemed to be related to protocol treatment are included. Patients aged 60 years or younger who served as a younger reference group for the pharmacokinetic study are excluded
Measure: Number; unit: Participants
Groups:
- Paclitaxel + Gemcitabine: Patients received 1000 mg /m^2 of gemcitabine on Day 1 and 8 and 175 mg/m^2 of paclitaxel on Day 1 intravenously every 21 days for 6 cycles ( 1 cycle = 21 days)
Arm/Group | Paclitaxel + Gemcitabine
Number analyzed (Participants) | 51
Participants
  Abdominal pain/cramping | 2
  Acidosis | 1
  Allergic reaction | 1
  Anemia | 6
  Anorexia | 3
  Bone pain | 1
  Cardiac ischemia/infarction | 1
  Chest pain,not cardio or pleur | 1
  Confusion | 1
  Constipation/bowel obstruction | 2
  Creatinine increase | 1
  Dehydration | 1
  Diarrhea without colostomy | 1
  Dizziness/light headedness | 1
  Dyspepsia/heartburn | 1
  Dyspnea | 6
  Edema | 1
  Fatigue/malaise/lethargy | 8
  Febrile neutropenia | 1
  Gastric ulcer | 1
  Hyperglycemia | 3
  Hyperkalemia | 2
  Hypotension | 2
  Infection w/o 3-4 neutropenia | 1
  Infection with 3-4 neutropenia | 3
  Infection, unk ANC | 1
  Leukopenia | 6
  Muscle weakness (not neuro) | 1
  Myalgia/arthralgia, NOS | 1
  Nausea | 3
  Neuropathic pain | 1
  Neutropenia/granulocytopenia | 26
  PRBC transfusion | 10
  Pain-other | 3
  Pleural effusions | 1
  Pneumonitis/infiltrates | 1
  Renal failure | 1
  Respiratory infect w/ neutrop | 1
  SGOT (AST) increase | 1
  Sensory neuropathy | 3
  Supraventricular arrhythmia | 1
  Thrombocytopenia | 2
  Thrombosis/embolism | 2
  Urinary tr infect w/ neutrop | 2
  Urinary tr infect w/o neutrop | 2
  Ventricular arrhythmia | 2
  Vomiting | 1
  Weakness (motor neuropathy) | 2

5. Primary Outcome: Determine the Feasibility of Accruing Patients With Metastatic Bladder Cancer Who Are 70 and Older to Chemotherapy Protocols
Description: Sixty patients aged 70 years and older were to be accrued to the study. The feasibility of accrual was determined that accrual of 3 patients per month in the age 70 and older range would allow for an expeditiously conducted phase II trial. If, after a 3 month start-up period, 3 or more patients aged 70 years and older were accrued per month for the duration of the trial, it was deemed reasonable to consider further trials in this elderly population.
Time Frame: 66 months (protocol activated on 7/1/2001 and closed to accrual on 12/15/2006)
Population: A total of 55 patients aged 70 years and older were registered to this protocol from July, 2001 to December, 2006.
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Gemcitabine (Elderly Cohort: Age >= 70)
Number analyzed (Participants) | 55
participants | 55

6. Secondary Outcome: Feasibility of Patient-reported Outcome Measures for Patients Aged 70 Years and Older: Form Submission Rate
Description: Patients were required to complete three self-administered questionnaires at entry, prior to the administration of any cytotoxic therapy: the Medical Conditions Questionnaire, Instrumental Activities of Daily Living Form that evaluates functional status, and the Feelings Questionnaire that evaluates depression status. Feasibility is defined in four ways: 1) submission rates for each of three patient self-administered questionnaires (> 60%); 2) the number of items missing within each scale (< 5%); 3) a description of the level of assistance required for self-administration of the questionnaires; and 4) the average amount of time it takes patients to complete each of the three questionnaires. Level of assistance is defined as the need to 1) read the questionnaire to the patient, 2) explain the meaning of items, 3) explain the response format, and 4) complete the questionnaire for the patient; an other category of assistance will be included.
Time Frame: at study entry (prior to administration of any treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel + Gemcitabine (Elderly Cohort: Age >= 70)
Number analyzed (Participants) | 51
percentage of participants
  Medical Conditions Questionnaire | 98
  Instrumental Activities of Daily Living Form | 98
  Feelings Questionnaire | 98

7. Secondary Outcome: Feasibility of Patient-reported Outcome Measures for Patients Aged 70 Years and Older: Median Time of Complete Forms
Description: Patients were required to complete three self-administered questionnaires at entry, prior to the administration of any cytotoxic therapy: the Medical Conditions Questionnaire, Instrumental Activities of Daily Living Form that evaluates functional status, and the Feelings Questionnaire that evaluates depression status. Feasibility is defined in four ways: 1) submission rates for the each of three patient self-administered questionnaires (> 60%); 2) the number of items missing within each scale (< 5%); 3) a description of the level of assistance required for self-administration of the questionnaires; and 4) the average amount of time it takes patients to complete each of the three questionnaires. Level of assistance is defined as the need to 1) read the questionnaire to the patient, 2) explain the meaning of items, 3) explain the response format, and 4) complete the questionnaire for the patient; an other category of assistance will be included.
Time Frame: at study entry (prior to administration of any treatment)
Population: Eligible patients aged 70 years and older who had received any treatment were included in the analysis. One non-compliant patient who did not complete any of the forms was excluded. Patients aged 60 years or younger who served as a younger reference group for the pharmacokinetic study were excluded from analysis.
Measure: Median (Full Range); unit: minutes
Arm/Group | Paclitaxel + Gemcitabine (Elderly Cohort: Age >= 70)
Number analyzed (Participants) | 50
minutes
  Medical Conditions Questionnaire | 5 [1 to 45]
  Instrumental Activities of Daily Living Form | 3 [1 to 45]
  Feelings Questionnaire | 2 [1 to 30]

8. Secondary Outcome: Assess the Feasibility of Patient-reported Outcome Measures for Patients Aged 70 Years and Older: at Least One Type of Assistance Required
Description: Patients were required to complete three self-administered questionnaires at entry, prior to the administration of any cytotoxic therapy: the Medical Conditions Questionnaire, Instrumental Activities of Daily Living Form that evaluates functional status, and the Feelings Questionnaire that evaluates depression status. Feasibility is defined in four ways: 1) submission rates for the three patient self-administered questionnaires (> 60%); 2) the number of items missing within each scale (< 5%); 3) a description of the level of assistance required for self-administration of the questionnaires; and 4) the average amount of time it takes patients to complete each of the three questionnaires. Level of assistance is defined as the need to 1) read the questionnaire to the patient, 2) explain the meaning of items, 3) explain the response format, and 4) complete the questionnaire for the patient; an other category of assistance will be included.
Time Frame: at study entry (prior to administration of any treatment)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel + Gemcitabine (Elderly Cohort: Age >= 70)
Number analyzed (Participants) | 50
percentage of participants
  Medical Conditions Questionnaire | 28
  Instrumental Activities of Daily Living Form | 42
  Feelings Questionnaire | 34

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events weekly after protocol treatment for cycle 1 (1 cycle = 21 days) and then weekly for the first 2 weeks of protocol treatment for cycle 2-6 and after completion of protocol treatment.
Description: Elderly Cohort (Age >= 70 years)
Arm/Group | Paclitaxel + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 5/51
Other Adverse Events (participants affected / at risk) | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel + Gemcitabine (N=51)
Cardiovascular-other (Cardiac disorders) | 1
Supraventricular arrhythmia (Cardiac disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Flu-like symptoms-other (General disorders) | 1
Reportable adverse event, NOS (General disorders) | 2
Respiratory infect w/ neutrop (Infections and infestations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel + Gemcitabine (N=51)
Anemia (Blood and lymphatic system disorders) | 29
PRBC transfusion (Blood and lymphatic system disorders) | 10
Blurred vision (Eye disorders) | 4
Abdominal pain/cramping (Gastrointestinal disorders) | 6
Constipation/bowel obstruction (Gastrointestinal disorders) | 16
Diarrhea without colostomy (Gastrointestinal disorders) | 12
Esophagitis/dysphagia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 25
Stomatitis/pharyngitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 9
Edema (General disorders) | 14
Fatigue/malaise/lethargy (General disorders) | 42
Fever without neutropenia (General disorders) | 8
Pain-other (General disorders) | 8
Rigors/chills (General disorders) | 6
Sweating (General disorders) | 4
Allergic reaction (Immune system disorders) | 3
Infection with 3-4 neutropenia (Infections and infestations) | 3
Urinary tr infect w/o neutrop (Infections and infestations) | 4
Alkaline phosphatase increase (Investigations) | 8
Creatinine increase (Investigations) | 7
Leukopenia (Investigations) | 12
Neutropenia/granulocytopenia (Investigations) | 36
SGOT (AST) increase (Investigations) | 11
SGPT (ALT) increase (Investigations) | 4
Thrombocytopenia (Investigations) | 20
Weight loss (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 23
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 20
Dizziness/light headedness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 5
Neuropathic pain (Nervous system disorders) | 4
Sensory neuropathy (Nervous system disorders) | 21
Taste disturbance (Nervous system disorders) | 4
Weakness (motor neuropathy) (Nervous system disorders) | 5
Confusion (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 12
Urinary frequency/urgency (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 27
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No